CLINICAL TRIAL: NCT03544723
Title: A Phase 2, Multi-Center, Open Label Study to Evaluate Adenoviral p53 (Ad-p53) in Combination With Immune Checkpoint Inhibitor Therapy in Patients With Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma and Other Tumors Approved for Anti-PD-1 or Anti-PD-L1 Therapy
Brief Title: Safety and Efficacy of p53 Gene Therapy Combined With Immune Checkpoint Inhibitors in Solid Tumors.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: MultiVir, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ad-p53-002
Record Dates: First submitted 2018-05-09; First posted 2018-06-04 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Solid Tumor; Lymphoma
Keywords: immune checkpoint inhibitor; anti-PD-1; anti-PD-L1; immune therapy; squamous cell cancer; solid tumor; lymphoma; carcinoma; breast cancer triple negative; cervical cancer; gastric cancer; gastroesophageal junction cancer; esophageal cancer; head and neck squamous cell cancer; hepatocellular cancer; Hodgkin's disease; non-small cell lung cancer; small cell lung cancer; melanoma; merkel cell cancer; MSI-H/dMMR; renal cell carcinoma; urothelial carcinoma; gene therapy; p53 tumor suppressor
MeSH Terms: conditions — Lymphoma; Neoplasms, Squamous Cell; Carcinoma; Triple Negative Breast Neoplasms; Uterine Cervical Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Liver Neoplasms; Hodgkin Disease; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Melanoma; Carcinoma, Merkel Cell; Carcinoma, Renal Cell; Carcinoma, Transitional Cell | interventions — advexin; Nivolumab; pembrolizumab; atezolizumab; durvalumab

STUDY DESIGN:
Intervention Model Description: Intratumoral Ad-p53 combined with approved immune checkpoint inhibitor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ad-p53 with anti-PD-1/anti-PD-L1 100% of patients (Experimental): Up to 40 patients, all patients treated with intra-tumoral Ad-p53 (dose determined by tumor size) in combination with IV physician's choice of approved immune checkpoint inhibitor
  Interventions: Drug: Ad-p53

INTERVENTIONS:
Drug: Ad-p53 — Antineoplastic, Monoclonal Antibody; PD-1/PD-L1 Inhibitors. Immunotherapy. Gene Therapy.
  Other Names: anti-PD-1/anti-PD-L1; nivolumab; pembrolizumab; atezolizumab; durvalumab

SUMMARY:
This is a single arm Phase 2 study of the combination of adenoviral p53 (Ad-p53) gene therapy administered intra-tumorally with approved immune checkpoint inhibitors in patients with recurrent or metastatic cancers. Comparison will be made to historical data. General safety and efficacy using RECIST 1.1 and Immune-Related Response Criteria as well as ECOG performance will be utilized.

DETAILED DESCRIPTION:
This is a Phase 2 study of the combination of Ad-p53 administered intra-tumorally in combination with physician's choice of FDA approved immune checkpoint inhibitor therapy in patients with recurrent or metastatic cancers. This is a safety and efficacy study with a single cohort, consisting of the combination of Ad-p53 and infusions of immune checkpoint inhibitors. Immune checkpoint inhibitor treatments will be administered in accordance with FDA package inserts. Comparison will be made to historical data. General safety and preliminary efficacy will be determined using RECIST 1.1, ECOG status and Immune-Related Response Criteria. Biomarker testing of archival or fresh tissue is performed during the study. Enrollment will be up to 40 patients.

ELIGIBILITY:
Inclusion Criteria

1. Signed informed consent.
2. Male or female greater than or equal to 18 years of age (females of childbearing potential must be non-pregnant with a negative pregnancy test and non-lactating). Males and females must use contraception for the duration of the study.
3. Primary diagnosis must be histologically confirmed.
4. Progression or Recurrence of solid tumors or lymphoma suitable for anti-PD-1/anti-PD-L1 therapy.
5. As far as possible, all target lesions utilized for RECIST response determination should be suitable for ultra-sound, CT or endoscopic guided intra-tumoral injection. If all target lesions cannot be treated with Ad-p53, but the patient is otherwise suitable for the study, this should be reviewed with the Sponsor.
6. Patients entered on the study must have disease that that is evaluable for response using RECIST 1.1 criteria with a minimum measurable lesion size of the longest axis greater than or equal to 1.0 cm (CT/MRI) or greater than or equal to 2.0 cm (non-helical CT), or nodal shortest diameter greater than or equal to 1.5 cm by CT/MRI.
7. No brain metastases or treated and stable brain metastases
8. ECOG Performance Status 0-1
9. Life expectancy greater than or equal to 6 months.
10. Adequate bone marrow and hepatic function as evidenced by the following:

    1. ANC greater than or equal to 1500 cells/mm3
    2. AST/SGOT and/or ALT/SGPT less than or equal to 3.0 x ULN
    3. Alkaline phosphatase less than or equal to 5 x ULN
    4. Platelet count greater than or equal to 100,000 cells/mm3
    5. Hemoglobin ≥9.0 g/dL
    6. Creatinine less than 2.0 mg/dL or creatinine clearance greater than or equal to 50 mL/min
    7. Total bilirubin less than 1.5 x ULN
    8. Serum albumin greater than or equal to 3.0 g/dL
11. Favorable tumor p53 biomarker profile as defined by wild type p53 gene sequence, or less than 20 percent p53 positive tumor cells by immunohistochemistry (IHC), or p53 gene mutations that will not inhibit normal p53 function such as gene deletions, truncations, or frame-shift mutations that result in non-functional p53 tetramerization. Mutant p53 gene profiles should be reviewed with the Sponsor to confirm eligibility.
12. Normal troponin blood levels.
13. Echo with normal ejection fractions.
14. QTcb less than or equal to 470 ms
15. Normal lung oxygen saturation by pulse oximeter.
16. Coagulation status should be suitable for intra-tumoral injections. Prothrombin Time (PT) less than or equal to 1.5 x ULN (or INR less than or equal to 1.3)*, Partial thromboplastin time (PTT) less than or equal to 1.5 x ULN* *Prolongation in INR, PT, and PTT when the result is from therapeutic anti-coagulation treatment are permitted for patients whose injectable lesions are cutaneous and/or subcutaneous such that direct pressure could be applied in the event of excessive bleeding.

Exclusion Criteria

1. History of allergic reactions to any components of the treatments (Ad-p53 or immune checkpoint inhibitors).
2. Active alcohol dependence
3. Neuropathy of less than or equal to grade 2 CTCAE.
4. Except for ongoing treatment with anti-PD-1 or anti-PD-L1 which is permitted (see Inclusion Criterion #4 above), there should be no other antibody-based therapy, targeted small-molecule therapy, hormonal therapy, chemotherapy, radiation, biological or investigational therapy within 14 days of first administration of Study Treatment (C1D1). Subjects with prior cytotoxic or investigational products less than 2 weeks prior to trial treatment might be eligible after discussion between investigator and Sponsor, if toxicities from the prior treatment have been resolved to Grade 1 (NCI CTCAE). If a patient with HNSCC is receiving combination pembrolizumab plus chemotherapy, the first Ad-p53 Study Treatment should be administered 2 weeks following the completion of final chemotherapy treatments and 5 days before their next anti-PD-1/anti-PD-L1 scheduled dose. Ad-p53 intratumoral injections should not be given within 24 hours of immune checkpoint inhibitor infusions.
5. Prior additional malignancy within 2 years except for non-melanoma skin cancer, carcinoma in situ of the breast, oral cavity, cervix or other cancers, unless approved by the Sponsor.
6. Prior autologous or allogenic organ or tissue transplantation.
7. Severe, active comorbidity, including any of the following:

   1. Active clinically serious infection (grade 2 or greater, CTCAE) or requiring intravenous antibiotics at the time of study treatment.
   2. Thrombotic or embolic event within the last 6 months unless approved by the Sponsor.
   3. Bleeding or evidence or history of clinically significant bleeding diathesis or coagulopathy within the last 3 months
   4. Uncontrolled hypertension despite treatment with anti-hypertensive medication (systolic blood pressure less than160 mmHg or diastolic blood pressure less than 100 mmHg)
   5. Must not have active, known or suspected autoimmune disease or be immunosuppressed
   6. Known acute or chronic hepatitis B or hepatitis C infection with signs of immunosuppression
   7. Known significant immunodeficiency due to underlying illness (e.g. HIV/AIDS) and/or immunosuppressive medication including high-dose corticosteroids; HIV patients may be approved by the Sponsor if on treatment with appropriate viral titers.
   8. Severe bleeding, hemoptysis, gastrointestinal hemorrhage, CNS bleeding, clinically significant hemorrhage or vaginal bleeding during the last 6 months
   9. Active brain metastases or leptomeningeal metastases are not allowed
   10. Subjects must not have evidence of autoimmune pneumonitis or inflammatory lung disease on CT scan and chest x-ray. Pneumonitis secondary to radiation scarring is permitted in the absence of dyspnea.
8. QTCb less than 470 ms
9. Systemic corticosteroid treatment for more than 6 months at doses above 10 mg prednisolone or equivalent before study entry
10. Psychological, familial, sociological or geographical or other condition which in the opinion of the investigator would not permit study follow-up or other compliance with the study protocol.
11. Subjects may not have target tumors for Ad-p53 injection adjacent to vital structures such as carotid arteries.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy endpoint is objective response rate (ORR) | Change in tumor size at the end of Cycle 2 (each cycle is 28 days)
  Objective response rate will be evaluated by RECIST 1.1
Safety assessments of adverse events per CTCAE | Signed Informed Consent through 30 Days following the final treatment
  Safety evaluations will tabulate adverse events per CTCAE

SECONDARY OUTCOMES:
Preliminary assessment of Duration of Response (DoR) by RECIST 1.1 | Day 1 through end of study, approximately 2 years
  RECIST 1.1 will be used to determine Duration of Response (DoR)
Preliminary assessment of progression free survival (PFS) by RECIST 1.1 | Day 1 through end of study, approximately 2 years
  RECIST 1.1 will be used to determine progression free survival

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Robert H. Lurie Comprehensive Cancer Center | Northwestern University, Chicago, Illinois
  - Rush University Cancer Center, Chicago, Illinois
  - Morristown Medical Center, Morristown, New Jersey

IPD SHARING:
Plan to Share IPD: No
Journal articles and posters, no identifiable data